CLINICAL TRIAL: NCT06337994
Title: Treatment of Post-traumatic Cognitive Dysfunction With Memantine Hydrochloride, an N-methyl-D-aspartate (NMDA)-Type Receptor Blocker: a Clinical Trial
Brief Title: Memantine Hydrochloride for Treatment of Cognitive Dysfunction Due to Traumatic Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherifa Ahmed Hamed, Professor of Neurology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUH-Neurol-TBI_2024
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Treatment of Cognitive Deficits After Traumatic Brain Injury
Keywords: Traumatic brain injury; closed head injury; cognition; memory; N-methyl-D-aspartate (NMDA)-type receptors; NMDA blocker; memantine hydrochloride
MeSH Terms: conditions — Brain Injuries, Traumatic; Head Injuries, Closed | interventions — Memantine

STUDY DESIGN:
Intervention Model Description: parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug treatment (interventional) (Active Comparator): - number of participant: >/= 60. This open-label clinical trial consisted of 24 weeks of memantine intake period, followed by 4-week (or more) post-trial observation period to monitor the drug adverse effects (e.g. sleep problems, sleepiness, sedation, anxiety, weight change and hypotension). Clinic visits will be scheduled at baseline and follow-ups after 6, 12, 18, 24 weeks of treatment initiation. Concomitant medications were essentially kept unchanged during the trial, i.e. the intake of antidepressant or antianxiologic psychotropic medications, psychotherapy to treat depressive or anxiety symptoms does not exclude participation in the study.
  Memantine was added to each patient's current medication, with the initial dosage of 5 mg/day (once daily). The dosage was then increased to 10 mg/day after a week and maintained till the end of the study. In the case of intolerance to this increase, the dosage was flexibly adjusted according to the condition of the patient.
  Interventions: Drug: Memantine Hydrochloride
- No intervention (No Intervention): number of participants: >/= 40

INTERVENTIONS:
Drug: Memantine Hydrochloride — Memantine was added to each patient's current medication, with the initial dosage of 5 mg/day (once daily). The dosage was then increased to 10 mg/day after a week and maintained till the end of the study. In the case of intolerance to this increase, the dosage was flexibly adjusted according to the condition of the patient.
  Other Names: Active arm
  Arms: Drug treatment (interventional)

SUMMARY:
Posttraumatic consequences are common causes of disability and long-term morbidity. They include cognitive dysfunction, seizures, headache, dizziness, fatigue, sensory deficits, neurodegeneration and psychiatric disorders (e.g. posttraumatic stress disorder, depression, anxiety, etc). Diffuse axonal injury and disruption of normal neuronal function are the most common and important pathologic features of traumatic primary closed head injury. depression, anxiety, etc). Excitotoxicity and apoptosis caused by activation of N-methyl-D-aspartate (NMDA) glutamate receptors, are two main suggested mechanisms of traumatic neuronal cell death and posttraumtic neurologic adverse consequences. Experimental and clinical studies have demonstrated that memantine hydrochloride, NMDA-type glutamate receptor antagonist, could have beneficial effect in treatment of posttraumatic cognitive dysfunction. Memantine may contribute to cognitive improvements in TBI by decreasing the synaptic 'noise' resulting from excessive NMDA receptor activation, inhibition of β-amyloid mediated toxicity and readjustment of the balance between inhibition and excitation on neuronal networks in the central nervous system (CNS).

DETAILED DESCRIPTION:
Posttraumatic consequences are common causes of disability and long-term morbidity. Traumatic brain injuries (TBIs) are traditionally classified into primary and secondary injuries. Primary brain injury is usually mechanically induced and occurs at the moment of injury while secondary injury is not mechanically induced, delayed from the moment of injury and may superimpose a previously injured brain by mechanical forces. Primary brain injury may be associated with focal scalp injury, skull fractures, brain contusion caused by contact (i.e. an object striking the head or the brain striking the inside of the skull) as well as diffuse axonal brain injury which is usually caused by acceleration-deceleration forces or rotational acceleration of the brain as a result of unrestricted movement of the head, shearing and tensile forces and compressive strains. Diffuse axonal injury and disruption of normal neuronal function are the most common and important pathologic features of TBI. The latter is mostly microscopic damage and is often not visible in neuroimaging. Consequences of TBI include cognitive dysfunction, seizures, headache, dizziness, fatigue, sensory deficits, neurodegeneration and psychiatric disorders (e.g. posttraumatic stress disorder, depression, anxiety, etc). Excitotoxicity and apoptosis are two main suggested mechanisms of traumatic neuronal cell death. The N-methyl-D-aspartate (NMDA) glutamate receptors are implicated in these mechanisms. Furthermore, the activation of NMDA receptors by glutamate promotes the production of reactive oxygen species (ROS) and nitric oxide (NO) which further exacerbate secondary cell injury. NMDA receptor plays a pivotal role in learning and memory. Experimental and clinical studies have demonstrated that memantine hydrochloride, NMDA-type glutamate receptor antagonist, could have beneficial effect in treatment of posttraumatic cognitive dysfunction. Memantine is an FDA-approved drug for the treatment of moderate to severe Alzheimer's disease and is also used clinically for the treatment of some patients with Parkinson's disease. Memantine is effective in blocking excessive activity of NMDA-type glutamate receptors and reduces the progression of dementia. Memantine has shown to be neuroprotective in animal models of cerebral and spinal cord ischemia and in models of TBI. Memantine may contribute to cognitive improvements in TBI by decreasing the synaptic 'noise' resulting from excessive NMDA receptor activation, inhibition of β-amyloid mediated toxicity and readjustment of the balance between inhibition and excitation on neuronal networks in the CNS. It showed beneficial effects in treating post-injury synaptic dysfunction in the neocortex, partially reversing deficits in long-term potentiation (LTP), mitigating pathologic NMDAR loss, and reducing tau phosphorylation and β-amyloid expression. Memantine spares hippocampal neurons after a single moderate/severe or repetitive TBI and normalizes LTP, β-amyloid and tau expressions, and neuroinflammation abnormalities in a repeat experimental model of TBI. In rodent studies, memantine dramatically increased adult hippocampal neurogenesis. Memantine does not have the significant negative side effects, such as hallucinations and coma of other NMDAR antagonists. High doses (≥20 mg/d) may cause non-serious side effects, e.g. dizziness, anxiety, restlessness or agitation,

ELIGIBILITY:
Inclusion Criteria:

* Adults (age: 18 - 60 years old)
* History of primary traumatic closed head injury
* At least 6 months after TBI
* Mild/moderate previous TBI
* Normal neuroimaging of the brain at the period of the study.

Exclusion Criteria:

* Secondary injury or superimpose injury on a brain already affected by a mechanical injury
* patients with duration of illness less than 6 months
* History of open or severe head injuries
* Severe neurologic consequences after TBI
* Post traumatic seizures
* Posttraumatic hydrocephalus'
* Posttraumatic abnormal neuroimaging of the brain
* History of chronic mental or neurologic disorders (e.g. comorbid schizophrenia, severe manic phase of bipolar disorder or intellectual disability).
* Substance abuse
* Pregnancy
* Individuals with the following physical conditions that are described in manufacturer's package including history of epilepsy or convulsion, renal dysfunction, factors increasing urine pH and severe liver dysfunction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The severity of traumatic brain injury (TBI) | Baseline
  (1) The severity of TBI at onset which was assessed according to (a) Glasgow coma scale (GCS) determined at the time of injury. (b)The duration of loss of consciousness (LOC) at the time of injury: (c) The time elapsed from injury to the moment when patients can demonstrate continuous memory of what is happening around them (i.e. orientation).
The symptoms of depression | Baseline
  (2) Beck's Depression Inventory - II (BDI-II)
The symptoms of anxiety | baseline
  (3) Hamilton Anxiety Rating Scale (HAM-A):
The cognitive function | baseline
  The validated versions of Mini-Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA) will be used to assess cognition. Each takes ~10-15 min to be administered.

SECONDARY OUTCOMES:
Quality of life after drug treatment | 8, 16, and 24 weeks
  (1) The brief WHO quality of life questionnaire (WHOQOL-brief) will be used for assessment. WHO defines Quality of Life as an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns.
Re-evaluation of the cognitive function after drug treatment | 8, 16, and 24 weeks
  The validated versions of Mini-Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA) were used to assess cognition as described above.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Faculty of Medicine, Hospital of Neurology, Psychiatry and Neurosurgery, Asyut, Egypt

REFERENCES:
- [Background] Bramlett HM, Dietrich WD. Long-Term Consequences of Traumatic Brain Injury: Current Status of Potential Mechanisms of Injury and Neurological Outcomes. J Neurotrauma. 2015 Dec 1;32(23):1834-48. doi: 10.1089/neu.2014.3352. Epub 2014 Dec 19. PMID 25158206
- [Background] Guerriero RM, Giza CC, Rotenberg A. Glutamate and GABA imbalance following traumatic brain injury. Curr Neurol Neurosci Rep. 2015 May;15(5):27. doi: 10.1007/s11910-015-0545-1. PMID 25796572
- [Background] Effgen GB, Morrison B 3rd. Memantine Reduced Cell Death, Astrogliosis, and Functional Deficits in an in vitro Model of Repetitive Mild Traumatic Brain Injury. J Neurotrauma. 2017 Feb 15;34(4):934-942. doi: 10.1089/neu.2016.4528. Epub 2016 Aug 8. PMID 27450515
- [Background] Chamoun R, Suki D, Gopinath SP, Goodman JC, Robertson C. Role of extracellular glutamate measured by cerebral microdialysis in severe traumatic brain injury. J Neurosurg. 2010 Sep;113(3):564-70. doi: 10.3171/2009.12.JNS09689. PMID 20113156
- [Background] Girouard H, Wang G, Gallo EF, Anrather J, Zhou P, Pickel VM, Iadecola C. NMDA receptor activation increases free radical production through nitric oxide and NOX2. J Neurosci. 2009 Feb 25;29(8):2545-52. doi: 10.1523/JNEUROSCI.0133-09.2009. PMID 19244529
- [Background] Sattler R, Xiong Z, Lu WY, Hafner M, MacDonald JF, Tymianski M. Specific coupling of NMDA receptor activation to nitric oxide neurotoxicity by PSD-95 protein. Science. 1999 Jun 11;284(5421):1845-8. doi: 10.1126/science.284.5421.1845. PMID 10364559
- [Background] Lipton SA. The molecular basis of memantine action in Alzheimer's disease and other neurologic disorders: low-affinity, uncompetitive antagonism. Curr Alzheimer Res. 2005 Apr;2(2):155-65. doi: 10.2174/1567205053585846. PMID 15974913
- [Background] Chen HS, Wang YF, Rayudu PV, Edgecomb P, Neill JC, Segal MM, Lipton SA, Jensen FE. Neuroprotective concentrations of the N-methyl-D-aspartate open-channel blocker memantine are effective without cytoplasmic vacuolation following post-ischemic administration and do not block maze learning or long-term potentiation. Neuroscience. 1998 Oct;86(4):1121-32. doi: 10.1016/s0306-4522(98)00163-8. PMID 9697119
- [Background] Dogan A, Eras MA, Rao VL, Dempsey RJ. Protective effects of memantine against ischemia-reperfusion injury in spontaneously hypertensive rats. Acta Neurochir (Wien). 1999;141(10):1107-13. doi: 10.1007/s007010050491. PMID 10550658
- [Background] Mei Z, Qiu J, Alcon S, Hashim J, Rotenberg A, Sun Y, Meehan WP 3rd, Mannix R. Memantine improves outcomes after repetitive traumatic brain injury. Behav Brain Res. 2018 Mar 15;340:195-204. doi: 10.1016/j.bbr.2017.04.017. Epub 2017 Apr 13. PMID 28412305